CLINICAL TRIAL: NCT07255872
Title: A Phase II/III Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of BL-M11D1 for Injection in Combination With Cytarabine + Daunorubicin or Venetoclax + Azacitidine in Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: A Study of BL-M11D1 in Combination With Cytarabine + Daunorubicin or Venetoclax + Azacitidine in Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M11D1-201
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Daunorubicin; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-M11D1 in Combination with Cytarabine + Daunorubicin or Venetoclax + Azacitidine (Experimental): Participants receive BL-M11D1 in Combination with Cytarabine + Daunorubicin or Venetoclax + Azacitidine for the first cycle (4 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M11D1; Drug: Cytarabine; Drug: Daunorubicin; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: BL-M11D1 — Administration by intravenous infusion for a cycle of 4 weeks.
Drug: Cytarabine — Administration in 4-week cycles.
Drug: Daunorubicin — Administration in 4-week cycles.
Drug: Venetoclax — Administration in 4-week cycles.
Drug: Azacitidine — Administration in 4-week cycles.

SUMMARY:
This study is an open, multicenter, dose-escalation and expansion, non-randomized phase II/III clinical trial to evaluate the safety, tolerability, pharmacokinetic characteristics, and preliminary efficacy of BL-M11D1 in combination with cytarabine + daunorubicin or venetoclax + azacitidine in patients with newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
The study cohorts include: Cohort A: Untreated newly diagnosed acute myeloid leukemia patients treated with BL-M11D1 in combination with cytarabine + daunorubicin. Cohort B: Untreated newly diagnosed acute myeloid leukemia patients treated with BL-M11D1 in combination with venetoclax + azacitidine.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. No gender restrictions;
3. Age: ≥18 years;
4. Expected survival time ≥3 months;
5. Newly diagnosed AML according to the World Health Organization (WHO) 2016 classification and confirmed by morphology;
6. ECOG performance status score ≤2;
7. Peripheral blood white blood cell count ≤25×10⁹/L before the first dose;
8. Organ function levels must meet the requirements;
9. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before starting treatment, and the serum/urine pregnancy test must be negative. Patients must not be breastfeeding; all enrolled patients (regardless of male or female) should adopt adequate barrier contraception throughout the entire treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Acute promyelocytic leukemia, acute transformation of chronic myeloid leukemia;
2. Previous treatment for AML;
3. Participation in other interventional or observational studies;
4. History of severe cardiovascular or cerebrovascular diseases within 6 months prior to screening;
5. Prolonged QT interval, complete left bundle branch block, third-degree atrioventricular block, frequent and uncontrollable arrhythmia;
6. Active autoimmune diseases and inflammatory diseases;
7. Diagnosis of other malignancies within 5 years prior to the first dose;
8. Poorly controlled hypertension;
9. Grade ≥3 lung disease as defined by CTCAE v5.0, history of interstitial lung disease requiring systemic steroid therapy, etc.;
10. Patients with central nervous system involvement;
11. Previous organ transplantation;
12. History of allergy to recombinant humanized antibodies or human-mouse chimeric antibodies, or allergy to any excipient component of BL-M11D1;
13. Positive human immunodeficiency virus antibody, active tuberculosis, active hepatitis B virus infection, or active hepatitis C virus infection;
14. Evidence of other clinically significant, poorly controlled infections requiring systemic treatment;
15. Clinically symptomatic or recurrent pleural, peritoneal, pelvic, or pericardial effusion requiring drainage;
16. Previous treatment with cytarabine, methylating agents, or investigational drugs for MDS;
17. Pregnant or lactating women;
18. Within 4 weeks prior to the first dose of the study drug, subjects must not have received any live vaccines or are not expected to receive live vaccines during the study participation;
19. Other conditions deemed by the investigator as unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Composite Response Rate（CRc） | Up to approximately 24 months
  CRc is defined as the proportion of patients who achieve any one of several pre-defined types of treatment response.
Phase IIa: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M11D1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BICR is defined as the time between the date subjects were randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Relapse-Free Survival (RFS) | Up to approximately 24 months
  Relapse-Free Survival (RFS) is defined as the time from randomization (or from the start of treatment for non-randomized studies) until the first occurrence of disease recurrence or death from any cause.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M11D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M11D1.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China